CLINICAL TRIAL: NCT00162552
Title: Clinical Trial of Pentoxifylline Administration Versus Placebo on Survival in Patients With Cirrhosis and Severe Liver Failure
Brief Title: Clinical Trial of Pentoxifylline in Patient With Cirrhosis
Acronym: PENTOCIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Saliha.DJANE, Delegation of clinical research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P030439; AOM03120
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2005-08

CONDITIONS: Cirrhosis; Liver Failure
Keywords: multicenter-randomized-trial; pentoxifyllinE; placebo; cirrhosis; liver failure; cytokine
MeSH Terms: conditions — Fibrosis; Liver Failure | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients with severe cirrhosis treated with Pentoxifylline
  Interventions: Drug: pentoxifylline
- 2 (Placebo Comparator): Patients with severe cirrhosis treated with a placebo
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: pentoxifylline — Patients with severe cirrhosis treated with Pentoxifylline
  Arms: 1
Drug: PLACEBO — Patients with severe cirrhosis treated with a placebo
  Arms: 2

SUMMARY:
In patients with cirrhosis and liver failure, pro-inflammatory cytokines (TNF alpha) might be responsible of severe complications and death. Thus, the prevention of cytokine production should prevent complications and mortality.

The aim of this study is to study the 2 months survival rate in patients with severe cirrhosis (Child-Pugh C) with pentoxifylline - an inhibitor of cytokine production. The 6 month mortality, the proportion of transplanted patients, the occurrence of complications (bacterial infection, renal failure, hepatic encephalopathy and gastrointestinal bleeding), plasma cytokine levels and fibrotest - a marker of fibrosis - will be also studied. This is a multicenter double blind randomized trial with a placebo.

All adult patients with severe cirrhosis might be randomized after written consent. Patients with severe carcinoma, intolerance or contraindication to pentoxifylline will not be included. Patients receive either pentoxifylline or placebo 3 times a day for 6 months. Three hundred and forty two patients are necessary to decrease mortality rate by 50% at 2 months in a beta risk of 10% and an alpha risk of 5%. Patients will be seen every month.

DETAILED DESCRIPTION:
The aim of this study is to study the 2 months survival rate in patients with severe cirrhosis (Child-Pugh C) with pentoxifylline - an inhibitor of cytokine production. The 6 month mortality, the proportion of transplanted patients, the occurrence of complications (bacterial infection, renal failure, hepatic encephalopathy and gastrointestinal bleeding), plasma cytokine levels and fibrotest - a marker of fibrosis - will be also studied. This is a multicenter double blind randomized trial with a placebo.

All adult patients with severe cirrhosis might be randomized after written consent. Patients with severe carcinoma, intolerance or contraindication to pentoxifylline will not be included. Patients receive either pentoxifylline or placebo 3 times a day for 6 months. Three hundred and forty two patients are necessary to decrease mortality rate by 50% at 2 months in a beta risk of 10% and an alpha risk of 5%. Patients will be seen every month.

ELIGIBILITY:
Inclusion Criteria:

* adult patient of more than 18 years
* child pugh C cirrhosis

Exclusion Criteria:

* pregnant woman
* Patient received anticoagulant
* Patient treated for arterial hypertension
* Patient with severe coronaropathy
* Patient with hyper sensibility of pentoxifylline
* Patient hospitalized for less 24 hours
* Patient admitted for a treatment of hepatocellular-carcinoma or COLLANGIO- carcinoma
* Patient with HIV
* Patient who has been transplanted
* Patient treated with immuno- suppressors
* Patient who has already received pentoxifylline for 3 months before inclusion
* Patient for whom the follow-up is considered impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2004-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
survival rate at 2 months | at 2 months

SECONDARY OUTCOMES:
- survival rate at 6 months | at six months
- Number of patient with liver transplantation | during the study
- Complications : bacterial infection, renal insufficiency, hepatic encephalopathy, gastrointestinal bleeding | during the study
- Fibrotest and Acutest before, at 2 months and at 6 months | at 2 months and at 6 months
- TNF alpha and IL6 plasma concentration before, at 2 months and at 6 months as predictive factor of mortality | at 2 months and at 6 months as predictive factor of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Didier LEBREC, MD, Principal Investigator — hopital Beaujon, APHP, france
Locations (1):
- Hôpital Beaujon, Clichy, France

REFERENCES:
- [Derived] Lebrec D, Thabut D, Oberti F, Perarnau JM, Condat B, Barraud H, Saliba F, Carbonell N, Renard P, Ramond MJ, Moreau R, Poynard T; Pentocir Group. Pentoxifylline does not decrease short-term mortality but does reduce complications in patients with advanced cirrhosis. Gastroenterology. 2010 May;138(5):1755-62. doi: 10.1053/j.gastro.2010.01.040. Epub 2010 Jan 25. PMID 20102716